CLINICAL TRIAL: NCT05160571
Title: A Retrospective Multicenter Review to Evaluate the Performance of the Ion Endoluminal System in Sampling Pulmonary Lesions
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-ION-R01
Record Dates: First submitted 2021-12-15; First posted 2021-12-16 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Lung Cancer; Pulmonary Nodule
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects with Ion Endoluminal sampling of pulmonary nodule: Subjects in which a pulmonary lesion biopsy was attempted or performed with the Ion Endoluminal System
  Interventions: Device: Ion Endoluminal System

INTERVENTIONS:
Device: Ion Endoluminal System — Ion Endoluminal Procedure for pulmonary nodule

SUMMARY:
This study is a retrospective multi-center chart review of patients who underwent an attempted biopsy of one or more pulmonary lesion(s) with the Ion Endoluminal System with the aim of assessing the overall performance of the system.

DETAILED DESCRIPTION:
This study is a retrospective multi-center chart review of patients who underwent an attempted biopsy of one or more pulmonary lesion(s) with the Ion Endoluminal System with the aim of assessing the overall performance of the system. The primary objectives of the study will be performance (evaluated by diagnostic yield and sensitivity for malignancy) and safety (assessed by rate of pneumothoraces and bleeding events).

ELIGIBILITY:
Inclusion Criteria:

* Subject was 18 years or older at the time of the procedure
* Biopsy procedure attempted/performed using the Ion Endoluminal System

Exclusion Criteria:

* Biopsy procedure was not attempted with the Ion Endoluminal System
* Biopsy procedure attempted with the Ion Endoluminal System occurred less than 12 months prior to IRB approval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who underwent an Ion Endoluminal Procedure with a pulmonary nodule, 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | Intra-operative through the one year follow up period
  Diagnostic yield of the sample obtained through the bronchoscopy procedure, with diagnostic yield defined as (true positives + true negatives)/(total number of lesions biopsied)
Sensitivity for malignancy | Intra-operative through the one year follow up period
  Sensitivity for malignancy of the sample obtained
Pneumothorax | Intra-operative
  Incidence of all pneumothoraces related to the Ion procedure
Bleeding | Intra-operative
  Incidence of bleeding in which an intervention was required, related to the Ion procedure. Interventions include: administration of cold saline, vasoactive substances, thrombin, or similar in response to active bleeding; use of bronchial/balloon blocker; use of bronchial artery embolization or resuscitation or ICU admission.

SECONDARY OUTCOMES:
Adverse events | Intra-operative through 30 days
  All adverse events related to the Ion procedure
Conversion to alternate approach or termination of procedure | Intra-operative
  Rate of procedures converted to an alternative approach or terminated. Conversion is defined as a change in the procedural approach (either a different technology [ex., electromagnetic navigational bronchoscopy] or a different procedure [ex., CT-guided transthoracic needle aspiration]) after the Ion catheter has entered the endotracheal tube. Termination is defined as prematurely ending the procedure after the Ion catheter has entered the endotracheal tube but before the biopsy sample has been obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Glen Bouder, MD, Principal Investigator — Winchester Medical Center
Locations (1):
- Winchester Medical Center, Winchester, Virginia, United States

IPD SHARING:
Plan to Share IPD: No